CLINICAL TRIAL: NCT06493318
Title: Evaluation of the Long-term Outcome of Dorsal Ligamentoplasty Reinforced With an Internal Brace in the Treatment of Scapholunate Instability
Acronym: ELIS
Status: Recruiting | Type: Observational
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-A00650-45
Record Dates: First submitted 2024-07-02; First posted 2024-07-09 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Wrist Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Dorsal ligamentoplasty reinforced with an internal brace — After a longitudinal dorsal incision of the wrist, an ECRB (extensor carpi radialis brevis) or palmaris longus hemi-tendon is harvested. The scapholunate positioning is adjusted using joystick pins. A 2.5 mm blind tunnel is made in the lunate and two 2.5 mm blind tunnels are made in the proximal and distal poles of the scaphoid. The tendon graft is threaded using a fiberloop and reinforced with suture tape. The graft is fixed in the proximal pole of the scaphoid with a swive-lock anchor (Arthrex®), then in the lunate, and finally fixed in the distal pole of the scaphoid by the same method. An anti-rotation scapho-capitate pin is then placed. This is maintained for 6 weeks during post-operative immobilization with a wrist orthosis. Rehabilitation begins after the pin is removed.

SUMMARY:
Prospective longitudinal multicenter observational cohort study conducted on a population of patients who underwent ligamentoplasty for scapholunate instability and agreed to be followed for a period of five years from the day of hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old who has been informed about the study and has not objected to the use of their personal data
* Patient who has undergone dorsal ligamentoplasty reinforced with an internal brace for scapholunate instability

Exclusion Criteria:

* Mental deficiency or any other reason that may interfere with understanding or strict application of the protocol
* Patient under legal protection, guardianship, or conservatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent ligamentoplasty for scapholunate instability
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2031-05-01 (Estimated); Study Completion 2031-05-01 (Estimated)

PRIMARY OUTCOMES:
Ligamentoplasty failure | Year 5
  Failure of the ligamentoplasty is defined by the need for secondary surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Monticelli - Vélodrome, Marseille, France